CLINICAL TRIAL: NCT05585385
Title: Effect of Backward Walking Versus Balance Training in Chronic Ankle Instability Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Ibrahim Ibrahim ElGayar, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003911
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Chronic Ankle Instability

STUDY DESIGN:
Intervention Model Description: Backward Walking Training and Balance Training
Who Masked: Participant, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Backward Walking Training (Experimental): The patients will receive BW training in addition to the traditional physical therapy program for 6 weeks.
  Interventions: Device: Backward Walking Training
- Balance Training (Experimental): The patients will receive balance training on the Biodex balance system in addition to the traditional physical therapy program for 6 weeks.
  Interventions: Device: Balance Training
- conventional treatment (Active Comparator): The patients will receive the traditional physical therapy program only for 6 weeks.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Device: Backward Walking Training — The subjects in this group will receive BW training program on an electric treadmill. The subject will be asked to walk, arms beside, in a backward manner on a level treadmill, zero inclination, with a warming up and cooling down period (5 minutes for each period). The subject walks at his self-selected and comfortable walking speed. A warm-up and cool-down period, in form of light jogging on a treadmill, will be done at speed of 1-2 m/sec. The total training is 30 minutes, three times a week for six consecutive weeks.
  Arms: Backward Walking Training
Device: Balance Training — Subjects in this group will receive balance training on Biodex Balance System for 3 sessions/ week, over 6 weeks period. Each subject will be instructed to stand with both legs on the "locked" platform. The researcher advances the platform to an unstable state while instructing the subject to focus on the visual feedback screen. Arms are free at the side of the body and not grasping handrails.
  After selecting the stability training program (dynamic balance training), Stability levels are changed depending on the subject's ability to maintain balance, and subjects are instructed to maintain their Center of Pressure (COP) in the smallest concentric rings (balance zones) of the Biodex Balance System monitor, named A zone.
  The stability level of the platform is set at level plate stability 8 (the most stable) for the first two sessions. After that, the plate stability is decreased by one level every two sessions to increase the difficulty in training.
  Arms: Balance Training
Other: Conventional treatment — Patients in this group will receive the traditional physical therapy program only for 3 sessions/ week, over 6 weeks period. The traditional physical therapy program is (evertors strengthening, short foot ex, heel raise ex, and calf stretch).
  Arms: conventional treatment

SUMMARY:
The goal of this clinical trial is to investigate the effect of backward walking versus balance training in patients with chronic ankle instability. The main question it aims to answer is:

Is there a difference between the effect of balance training and BW training on balance, ankle proprioception, risk of fall, and functional limitations in CAI patients?

DETAILED DESCRIPTION:
Lateral ankle sprains are among the most common musculoskeletal injuries. Approximately 40% of individuals who have ever suffered any lateral ankle sprain will develop chronic ankle instability which is defined as posterior mechanical and functional deficits in this joint.

Balance is the process that maintains the center of gravity within the body's support base, which needs constant adjustments with joint positioning and muscular activity. Many musculoskeletal and nervous system diseases can alter balance control. It has been reported that individuals with CAI have poor static and dynamic balance compared to those with normal ankles, and this affection of balance, increases the falling risks and leads to serious injuries.

A reversal of normal walking is simply recognized as retro-walking or backward walking (BW), where the toes first reach the ground and finish with the heel off. BW training causes changes in the motion control system and gait characteristics and exerts a positive effect on postural stability.

Sixty patients with chronic ankle instability will be assigned randomly into 3 equal groups; group A will receive BW training in addition to the traditional physical therapy program for 3 sessions/ week, over 6 weeks periods, Group B: will receive balance training on Biodex balance system in addition to the traditional physical therapy program for 3 sessions/ week, over 6 weeks periods, group C: will receive the traditional physical therapy program only for 3 sessions/ week, over 6 weeks periods.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects will complete a questionnaire by self-report (Cumberland Ankle Instability Tool (CAIT) to be characterized as having Functional Ankle Instability (FAI) ; All subjects' scores on CAIT will be less than 23 to be severely identified with FAI. Subjects will satisfy the following criteria:

   Having FAI that persists after the initial lateral ankle sprain and complaining of residual symptoms (repeated episodes of giving way or feeling of ankle joint instability) and suffering of repeating injury.
2. Having mechanical ankle instability on one ankle joint (will be identified by manual testing as talar tilt and anterior drawer test of the ankle to determine the integrity of ankle ligaments).
3. Their age ranges from 18 to 35 years.
4. Subjects with body mass index less than 30 kg/m2.
5. Not undergoing any formal or informal rehabilitation of the unstable ankle.

Exclusion Criteria:

1. Ankle joint swelling or any rheumatological disorders in both legs.
2. Ankle surgery in either leg.
3. Gross limitation in ankle range of motion in both legs.
4. Any joint disease or bony fracture in the lower extremity.
5. History of neurological disorder affecting the upper or lower extremities, vestibular dysfunction, or balance disorder.
6. Receiving formal or informal rehabilitation of their unstable ankle for 3 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Dynamic Balance Assessment | up to 6 weeks
  Dynamic balance is assessed by the Biodex stability system which has a high level of accuracy in determining dynamic equilibrium for postural control testing. It establishes three numeric stability indexes: Overall Stability Index (OSI), Anterior/Posterior Stability Index (APSI), and Medial/Lateral Stability Index (MLSI), to assess the body's deviation from its gravity center. The OSI indicates the overall score in all directions, while the APSI and MLSI represent the sagittal and frontal planes, respectively. The higher the stability, the lower the ranking.
Active repositioning accuracy of ankle joint | up to 6 weeks
  Ankle proprioception will be assessed by a digital goniometer. The starting position for ankle joint testing is 90 degree. The maximum ankle planter flexion for each subject will be measured, and half this max. range will be selected as the target position. Subjects will be asked to remain in that position for 10 seconds. The subject with closed eyes actively moves the ankle from starting position (90 degrees) to the targeted plantar-flexion angle with constant speed during the test (they were asked to return to the initial position and progressively move towards the target degree). This process would be repeated 3 times and the average error in active repositioning of the targeted angle would be taken.
Functional limitations | up to 6 weeks
  Functional disability will be assessed by the Foot and Ankle Disability Index (FAID).This index is a 34-item questionnaire divided into subscales, FADI and FADI sport. FADI contains 4 pain related items and 22 activity related items, while the FADI sport contains 8 activity related items. Each question can be scored on a 5- point Likert scale (from 0 to four). FADI and FADI sport are scored separately. FADI has total score of 104 points and FADI Sport 32 points. Both are transformed into percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Neveen A. Abdel Raoof, PhD, Study Chair — Cairo University; Ghada A. Abd Allah, PhD, Study Director — Cairo University; Rania R. Mohamed, PhD, Study Director — Cairo University; Amr A. Azzam, PhD, Study Director — National Institute of Neuromotor System
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Egypt